CLINICAL TRIAL: NCT06995235
Title: MAGenTA: Map of Tumor Genetic Actionability in Argentina
Brief Title: Map of Tumor Genetic Actionability in Argentina
Acronym: MaGenTA
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Hernan Garcia Rivello, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 3495
Record Dates: First submitted 2025-05-16; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms Malignant; Biomarkers
Keywords: panel genes; cancer patients; sequencing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Selection of clinically relevant case samples due to the frequency of the pathology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study of the human genome laid the foundations for the search for a large number of molecular alterations related to different diseases. The Precision medicine allows us to know molecular alterations that can be detected and targeted for therapeutic purposes. There is little data in Argentina about the incidence and frequencies of alterations molecules associated with the most frequent tumors. Through the selection of a gene panel, analysis of the genetic information obtained analysis allows classifying tumors from a point of view therapeutic. On the other hand, through the same panel, markers of resistance to drugs that allow the incorporation of retreatment therapies. Together with the proposed panel, the ancestry of the patients will be evaluated to determine whether the frequencies of molecular alterations vary between the different ethnic origins of the country.

DETAILED DESCRIPTION:
Platform Development A validation study of a new genetic panel of 52 genes will be carried out in tissue biopsies from adult subjects with the most prevalent solid tumors in Argentina.

In a first phase, 200 retrospective samples of different tumors and matrices (e.g. paraffin tissue, fine needle biopsy and fresh tumor) to be able to analytically validate the proposed panel. Reproducibility tests will be carried out, repeatability and determination of the detection limit for each of the 52 markers studied.

The choice of tumor types will be based on the frequency observed in the population from the Italian Hospital of Buenos Aires (HIBA), corroborated against agency data international cancer research (IARC-WHO). The distribution of samples of tumors (T) will be: 15% T digestive (colon), 15% T breast cancer, 15% T skin cancer (melanoma and basal cell carcinoma), 15% T lung cancer, 10% T prostate, 6% thyroid T, 6% ovarian T, 6% bladder/renal T and 12% rare T (nervous system central, musculoskeletal, head and neck, among others).

In a second phase, once fine-tuned and analytically validated, the panel will be available to the treating doctor who may request the panel with prior consent informed of the subject.

Tumor biopsies, both retrospective and prospective, are received and processed in the HIBA Pathological Anatomy Service by standardized methods that encompass embedding in paraffin (paraffin wad) and extraction of cellular genomic material (total cellular DNA -nuclear and mitochondrial- and RNA) by cutting 10 micron chips of thickness. Said paraffin material will be processed, in its entirety, with commercial kits of extraction of nucleic acids using Qiagen columns or equivalent.

Gene Panel Sample Study: Proposed Massive Sequencing Method

Thermo Fisher's S5 and Ion Torrent platforms will be used. The workflow comprises the amplification of specific regions and the generation of libraries to then be able to perform an emulsion PCR(Polymerase Chain Reaction). After a PCR enrichment step of emulsion, sequencing is carried out on chips of variable capacity, depending on the amount of data you wish to obtain. For the project, it is intended to process 32 samples in parallel with an Ion 540 chip.

To comply with international standards, a validation phase will be carried out gene panel according to the guidelines recently published by the College American Association of Pathologists and the American Genetics Association: "Guidelines for Validation of Next Generation Sequencing based on Oncology Panel. A Joint Consensus Recommendation of the Association for Molecular Pathology and College of American Pathologist", published in March 2017 6d

The Oncomine Focus Assay panel It is a multimarker analysis that is carried out in massive sequencing equipment (S5) that evaluates 52 genes associated with treatment of solid tumors for which there is scientific evidence of its usefulness diagnostic, prognostic and/or predictive of therapeutic response The system analyzes DNA and RNA extracted from the tumor piece -biopsy- or blood, for example. The catalog of detectable alterations includes 35 hotspot genes, 19 Copy Number Variations (CNVs) and 23 gene fusions.

ELIGIBILITY:
Inclusion Criteria:

Subjects 18 years of age or older Subjects diagnosed with cancer due to solid tumors who have a sample of tissue from a previous surgery or biopsy that is sufficient to be able to carry out the study methodology.

Subjects who agree to sign the informed consent

Exclusion Criteria:

Subjects who do not agree to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective samples of patients over 18 years of age from different tumors and matrices (e.g. paraffin tissue, fine needle biopsy and fresh tumor)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
massively parallel sequencing | 6 months
  Put into operation a massive gene sequencing platform second generation (massively parallel sequencing) for the development of a panel of precision genomic oncology in adult subjects diagnosed with solid tumors assisted at the Italian Hospital of Buenos Aires.

SECONDARY OUTCOMES:
Ancestry | 12 months
  Perform ancestry analysis in adult subjects diagnosed with solid tumors assisted at the Italian Hospital of Buenos Aires to determine the frequency of molecular alterations associated with these tumors according to the ethnic origin of the studied population.
Tumor genomic actionability map | 36 months
  Forge a tumor genomic actionability map in adult subjects with a diagnosis of solid tumors in Argentina, generating data on tumor frequencies and their associated molecular alterations that will be made available to the community medical and scientific throughout the country through a unified database.

CONTACTS AND LOCATIONS:
Overall Officials: Hernan Garcia Rivello, MD, Principal Investigator — Medical Doctor
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina